CLINICAL TRIAL: NCT01446718
Title: A Longitudinal Observational Cohort Study to Assess Sustained Immunogenicity up to 48 Months to Quadrivalent Human Papillomavirus Vaccine Among HIV-infected Girls and Boys Age 9-14 Years in Kenya
Brief Title: A Cohort Study to Assess Sustained Immunogenicity to qHPV Vaccine Among HIV-infected Girls and Boys Age 9-14 Years
Status: Completed | Type: Observational
Sponsor: Kenya Medical Research Institute (Other)
Collaborators: University of Washington (Other); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Nelly Rwamba Mugo, Dr., Kenya Medical Research Institute
Other Study IDs: (MISP)IISP 51802; NCT01998178 (obsolete NCT alias)
Record Dates: First submitted 2011-09-30; First posted 2011-10-05 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Human Papillomavirus; HIV-1 Infection
Keywords: quadrivalent vaccine; Human Papillomavirus
MeSH Terms: interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Plasma for HPV antibody testing there will be no long term sample storage
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Gardasil Vaccine: This is an extension of follow up for participants who received 3 doses of Gardasil vaccine in the "Immunogenicity and Safety of Quadrivalent Human Papillomavirus Vaccine in HIV-Infected Pre-Adolescent Girls and Boys in Kenya" study.
  Interventions: Biological: Gardasil vaccine

INTERVENTIONS:
Biological: Gardasil vaccine — 0.5ml of intramuscular vaccine in three doses
  Other Names: Gardasil

SUMMARY:
The purpose of this study is to determine sustained immunogenicity of the quadrivalent vaccine 'Gardasil', 48 months after initial vaccination, among HIV-1 infected boys and girls age 9-14 years. This age range is within the World Health Organization (WHO) stipulated guidelines for national programs for the vaccine.

DETAILED DESCRIPTION:
HIV-infected individuals bear a disproportionate disease burden of HPV-related diseases suggesting more rapid progression from HPV acquisition to malignancy. HIV infected women have a 2-22 fold increased risk for cervical cancer compared to uninfected women. The quadrivalent HPV vaccine marketed as "Gardasil" has demonstrated efficacy against type specific HPV infections known to cause 70% cervical cancer (HPV 16 & 18) and HPV 6 & 11 known to cause 90% of anogenital warts in populations of HIV negative young women.

Since the risk of HPV exposure persists throughout a person's sexual life, the duration of protection, especially when the vaccine is given in the pre-adolescent period, is critical to overall vaccine effectiveness. Extended follow up of HIV-uninfected individuals has shown sustained response to HPV vaccine for 8.4 and 6 years respectively to the bivalent and quadrivalent vaccines. However, other vaccines such as the hepatitis B vaccine have been shown to require additional dosages to be effective among HIV-infected persons.

Data on immunogenicity of the HPV vaccine among HIV infected adolescents is limited to a 12 month follow up period.

Current HPV vaccine guidelines target pre-sexual adolescents. Since the risk of HPV exposure persists throughout an individual's sexual life, the duration of protection provided by vaccination is critical to the overall vaccine effectiveness. Duration of sustained HPV 6/11/16/18 antibody response is directly related to vaccine effectiveness and determines the need for booster dosing.

The investigators therefore propose to extend follow up of 179 girls and boys in Kenya, age 9-14 years who have received 3 doses of the quadrivalent 'Gardasil' vaccine and assess for immunogenicity annually.

Study Location: Partners in Prevention, Thika site

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected
* age 9-14 years
* guardian/parental consent

Exclusion Criteria:

Participants will be excluded if they

* are severely ill as defined by Karnofsky <70
* have a diagnosis of malignancy
* on-going febrile illness (temperature ≥37.8°C), including active treatment for an opportunistic infection
* have received systemic corticosteroids within prior one year
* have received inactivated vaccine within prior 2 weeks, or live attenuated vaccine within prior 6 weeks
* have history of allergy to any products included in the HPV vaccine
* have received any of blood derivatives within prior 6 months
* are pregnant
* lack parental consent and/or parent declines to provide assent

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Study participants will be enrolled from the paediatric HIV-care clinic
Sampling Method: Non-Probability Sample
Enrollment: 179 (Actual)
Dates: Start 2014-12-15 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
immune response to vaccine specific HPV types | 48 months
  antibody response to HPV type 6, 11, 16, 18 measured by cLIA

SECONDARY OUTCOMES:
immune response to vaccine specific HPV types | 48 months
  HPV infection among sexually active HIV infected adolescents

CONTACTS AND LOCATIONS:
Overall Officials: Nelly R Mugo, MMed, MPH, Principal Investigator — Kenya Medical Research Institute